CLINICAL TRIAL: NCT01461954
Title: A Multi-Center, Randomized, Double-Masked Study to Evaluate the Clinical Efficacy and Safety of FST-100 Ophthalmic Suspension in the Treatment of Acute Viral Conjunctivitis
Brief Title: FST-100 in the Treatment of Acute Viral Conjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FST100-AVC-005
Record Dates: First submitted 2011-10-24; First posted 2011-10-28 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Acute Viral Conjunctivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FST-100 (Experimental)
  Interventions: Drug: FST-100
- FST-100 Vehicle (Placebo Comparator)
  Interventions: Drug: FST-100 Vehicle

INTERVENTIONS:
Drug: FST-100 — FST-100
  Arms: FST-100
Drug: FST-100 Vehicle — FST-100 Vehicle
  Arms: FST-100 Vehicle

SUMMARY:
This randomized, double masked, multi-center study is being conducted to support the safety and efficacy of FST-100 for the treatment of acute viral conjunctivitis. The study intends to show superiority of FST-100 ophthalmic suspension compared to vehicle for clinical resolution of acute viral conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of suspected acute viral conjunctivitis in at least one eye

Exclusion Criteria:

* Have a known sensitivity to any of the components of FST-100 or FST-100 vehicle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2013-05-17 (Actual); Primary Completion 2014-03-10 (Actual); Study Completion 2014-03-10 (Actual)

PRIMARY OUTCOMES:
Clinical resolution of acute viral conjunctivitis | 6-7 days

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (2):
- Ora Clinical Site, Andover, Massachusetts, United States
- Hospital São Paulo/Federal University of São Paulo (UNIFESP), São Paulo, Brazil